CLINICAL TRIAL: NCT07146152
Title: Empowering Women - Shared Decision-Making in Managing Cervical Precancer
Brief Title: Empowering Women - Shared Decision Making in Managing Cervical Precancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Region MidtJylland Denmark (Other); Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: EmpowerWomen2025
Record Dates: First submitted 2025-07-01; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: CIN2
Keywords: Shared decision making; Cervical precancer; Cervical intraepithelial neoplasia; Shared Decision-making; SDM; Patient Decision Aid; CIN2
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients with CIN2 recieving standard information about treatment choices (Standard of Care)
- Intervention Arm (Experimental): Patients with CIN2 receiving information about treatment options using a Patient Decision Aid to promote shared decision making.
  Interventions: Device: Patient Decision Aid

INTERVENTIONS:
Device: Patient Decision Aid — A Patient Decision Aid designed to help patients with CIN2 make informed decisions about wether they prefer operation (Loop Electrical Surgery) or active surveillance.
  Arms: Intervention Arm

SUMMARY:
The aim of this stepped-wedge randomized clinical trial is to assess the impact of implementing a patient decision aid during consultations with patients diagnosed with cervical precancer. Specifically, it will evaluate whether the decision aid enhances shared decision-making, improves the patient experience, and influences their treatment preferences.

The main questions this study aims to answer are:

1. Will the implementation of the patient decision aid increase the number of patients with cervical precancer who opt for surgery (loop electrical excision) compared to active surveillance?
2. Will the implementation of the patient decision aid improve patients' experience with the course of treatment for cervical precancer?

To evaluate this, researchers will compare patients receiving counseling with the support of the decision aid to those receiving standard counseling without the decision aid.

After the consultation, participants will complete questionnaires to share their experience. Data on treatment choices will be gathered from patient medical records.

ELIGIBILITY:
Inclusion criteria

* Newly diagnosed CIN2
* Age 18-50 years old

Exclusion criteria

* CIN2 or worse or conization surgery within the last 2 years.
* Pregnancy
* Immunosuppressed individuals, including those with HIV and organ transplant recipients
* Non-visible transformation zone
* Language difficulties requiring an interpreter or translator

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Surgical Intervention vs. Active Surveillance | The treatment decision will be documented immediately after it is made, expected within one month after inclusion.
  A comparison of the number of patients choosing surgical treatment during the study period.

SECONDARY OUTCOMES:
Decision Regret | From enrolment until 9 months follow-up.
  Decision regret will be measured using the validated "Decision Regret Scale", which ranges from 1 (indicating low regret) to 5 (indicating high regret).
Anxiety levels | From enrollment until 9 months follow-up.
  Participants' anxiety levels will be measured both before and after they make a decision regarding their treatment. The validated "State-Trait Anxiety Inventory" (STAI) will be used, which rates anxiety on a scale from 1 to 4, with 4 indicating the highest level of anxiety.
Shared decision making | Data will be collected from the time of inclusion and within a short period following the treatment decision, typically around 1 month after inclusion.
  Measurement of degree of shared decision-making from the participants' point of view using validated questionnaire "CollaboRATE". Patients report to which degree they felt the doctor fascilitated shared decision-making during the consultation. The scale ranges from 1 (to the lowest degree) to 9 (to the highest degree).
Shared Decision Making | Data will be collected from the time of inclusion and within a short period following the treatment decision, typically around 1 month after inclusion.
  The degree of shared decision-making will be assessed from the participants' point of view using the validated questionnaire "Shared Decision-Making Process-4".
Shared Decision Making | Data will be collected from the time of inclusion and within a short period following the treatment decision, typically around 1 month after inclusion.
  The extent of shared decision-making will be assessed from the participants' point of view using the validated questionnaire "Shared Decision Making Questionnaire Q9 (SDM-Q-9).
Shared Decision Making from the doctor's point of view. | Data will be collected at a single time point, immediately following the consultation in which the treatment decision is made.
  The degree of shared decision-making will be assessed from the physician's point of view using the validated questionnaire "Shared Decision Making Questionnaire - Physician Version".
Decisional conflict | The questionnaire is administered at two time points: prior to the consultation regarding treatment choice, and immediately after the consultation. Data collection is expected to be completed within one month of enrollment.
  Measurement of decisional conflict using the validated questionnaire "Decisional Conflict Scale". The scale ranges from 1 (low degree of decisional conflict) to 5 (high degree of decisional conflict).

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Hospital Gødstrup, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No